CLINICAL TRIAL: NCT02166320
Title: The Importance of Stent Design
Brief Title: Treatment of Malignant Strictures in Esophagus and Gastroesophageal Junction With Covered or Partially Covered Stent.
Acronym: StentMig
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Blekinge County Council Hospital (Other); Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/1034-31/3; 2009/1034-31/3 (Other: Ethical Review board, Karolinska Institute Stockholm)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Esophageal Cancer; Cancer of Gastro Esophageal Junction; Palliative Treatment
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Partially covered SEMS (Active Comparator): Boston Scientific Ultraflex SEMS
  Interventions: Device: Partially covered SEMS
- Fully covered SEMS (Experimental): Boston Scientific Wallflex Esophageal SEMS.
  Interventions: Device: Fully covered SEMS

INTERVENTIONS:
Device: Partially covered SEMS
  Arms: Partially covered SEMS
Device: Fully covered SEMS
  Arms: Fully covered SEMS

SUMMARY:
Self expandable stent (SEMS) constitutes the main palliative treatment in advanced esophageal cancer. The palliative effect of SEMS is immediate when it comes to relief of dysphagia. The duration of this effect is however questionable. The design of SEMS can be of importance since the device can dislodge and as a consequence of that dysphagia recur. The hypothesis has therefore been formulated that a partially covered SEMS is associated with less tendency to dislocate as compared to those SEMS, recently developed, which are covered through their entire length.

ELIGIBILITY:
Inclusion Criteria:

* Verified Squamous Cell Carcinoma or Adenocarcinoma of esophagus or Gastro Esophageal Junction (GEJ)
* Age above 18 years.
* Dysphagia scoring grade two or worse
* Not amenable for curative treatment
* Informed consent to participate

Exclusion Criteria:

* Concomitant cancer disease
* Inability to comply with study protocol
* Previous stent treatment
* Proximal location of the tumour in the esophagus.
* Need for more than one stent deployment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
SEMS dislocation in cm during first thirty days after stent insertion. | Thirty days from stent deployment.

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQOL) | Within three months of SEMS deployment.
Need for reintervention | Within three months after SEMS
Grade of dysphagia within three months of SEMS. | Three months after insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Johnsson, MdPhd, Principal Investigator — Sahlgrenska University Hospital, Clinic of Surgery; Magnus Nilsson, ass professor, Study Chair — Karolinska University Hospital
Locations (1):
- Erik Johnsson, Gothenburg, Sweden